CLINICAL TRIAL: NCT03564470
Title: An Open-Label, One-Arm, Multi-Site Trial of Precision Diagnosis Directing Target Total Therapy for Adult Ph-like Acute Lymphoblastic Leukemia
Brief Title: Precision Diagnosis Directing HDACi and TKI Target Therapy for Adult Ph-like ALL
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Hongsheng Zhou. M.D., Ph.D, M.D., Professor, Nanfang Hospital, Southern Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PDT-Ph-Like
Record Dates: First submitted 2018-06-09; First posted 2018-06-20 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Leukemia; Leukemia, Acute; Leukemia, Lymphoblastic; Leukemia, B-cell
Keywords: Acute Lymphoblastic Leukemia; Ph-like; Tyrosine Kinase Inhibitor; Histone Deacetylase Inhibitor
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, B-Cell | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chidamide (Experimental): Chidamide will be added to chidamide arm Ph-like ALL(CRLF2 high-expression, CRLF2/EPO/JAK2 rearrangement, JAK/IL-7R/SH2B3 mutation, etc).
  Interventions: Drug: Chidamide
- Dasatinib (Experimental): Dasatinib at a dose of 100mg/day will be added to Dasatinib arm of Ph-like ALL (CRKL high-expression, ABL1 or ABL2 or CSFR1 or PRGFRB rearrangement, etc).
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Chidamide — Chidamide will be administrated at dose of 10mg/day in chidamide arm in PDT-Ph-Like protocol. PDT-Ph-Like protocol for chidamide arm consists of diagnostic test (bone marrow aspiration, flow immunophenotyping, karyotyping，FISH, NGS, Flow-MRD), induction regimen (chidamide, prednisone, vincristine, cyclophosphamide, idarubicin, pegaspargase), consolidation regimen (chidamide, cytarabine, methotrexate, dexamethasone, cyclophosphamide, etoposide, 6-mercaptopurine, pegaspargase), MRD assessment and maintenance regimen, intrathecal injection chemotherapy, radiation therapy for CNS-involved leukemia and allogeneic hematopoietic stem cell transplantation.
  Other Names: HDACi chidamide
  Arms: Chidamide
Drug: Dasatinib — Dasatinib will be administrated at a dose of 100mg/day in dasatinib arm in PDT-Ph-Like protocol. PDT-Ph-Like protocol for dasatinib arm consists of diagnostic test (bone marrow aspiration, flow immunophenotyping, karyotyping，FISH, NGS, Flow-MRD), induction regimen (dasatinib, prednisone, vincristine, cyclophosphamide, idarubicin, pegaspargase), consolidation regimen (dasatinib, cytarabine, methotrexate, dexamethasone, cyclophosphamide, etoposide, 6-mercaptopurine, pegaspargase), MRD assessment and maintenance regimen, intrathecal injection chemotherapy, radiation therapy for CNS-involved leukemia and allogeneic hematopoietic stem cell transplantation.
  Other Names: TKI dasatinib
  Arms: Dasatinib

SUMMARY:
Ph-like ALL is a recently recognized high-risk subgroup and the optimal therapeutic approaches are poorly characterized. Based on the pediatric-inspired, PEG-L-asparaginase-intensified and MRD-directed PDT-ALL-2016 protocol, this open-label, two-arm, multi-site trial PDT-Ph-like-ALL is aimed to evaluate the safety and effect of oral histone deacetylase inhibitor chidamide and dasatinib for adult Ph-like ALL.

DETAILED DESCRIPTION:
Ph-like, or BCR-ABL1-like lymphoblastic leukemia is neoplasm of lymphoblasts committed to the B-cell lineage that lack the BCR-ABL1 translocation but show a pattern of the expression very similar to that seen in BCR-ABL1-positive ALL. Chidamide is a novel oral HDACi with promising activity in non-Hodgkin lymphoma (NHL). Based on the pediatric-inspired, PEG-L-asparaginase-intensified and MRD-directed PDT-ALL-2016 protocol, this open-label, two-arm, multi-site trial is aimed to evaluate the safety and effect of oral histone deacetylase inhibitor (HDACi) chidamide and tyrosine kinase inhibitor (TKI) dasatinib for adult Ph-like ALL/LBL. HDACi chidamide and TKI dasatinib will be added to chidamide and dasatinib group, respectively, from induction therapy to consolidation therapy (total courses of chidamide treatment: 5 courses for allo-HSCT after Consolidation Module-3; 12 courses for patients non-allo-HSCT after Consolidation Module 1-9). Primary study endpoint is event-free survival and secondary study endpoints are complete remission and MRD after induction, adverse event and overall survival.

Pretreatment: Dexamethasone, -3 to 0d;

Chidamide for chidamide arm: 10mg/d, po qd.

Dasatinib for Dasatinib arm: 100mg/d, po qd.

Induction:VCR: 1, 8, 15, 22; IDA: 1, 8; CTX: 1g/m2, 1; PEG-asp: 2000-2500IU/m2, 1, 15; Pred: 1-24;

MRD assessment: d14, 24, 45, and pre-allo-HSCT.

VLCAM (MRD1/d14>1%): CTX, d25; AraC 50mg/m2, d25-31, 26; 6-MP: 25-31, PEG-asp: 26;

Consolidation Module:

CM1: AraC 2g/m2, q12h, 1-2, Dex: 10mg/m2, 1-2, PEG-asp: 2, 6-MP: 1-7. IT: d1; CM2: MTX 3g/m2, 1, Dex: 10mg/m2, 1-2, PEG-asp: 2; 6-MP: 1-7; IT: d1; CM3: CTX 0.5g/m2, 1-3, PEG-asp: 2, 6-MP: 1-7, IT: d1.

Allo-HSCT: after CM3 when donors available. Non-HSCT: finish CM 4-9 and POMP maintenance.

CM4-6: repeat CM1-3. Re-Induction: after CM6. CM7-9: repeat CM1-3.

Maintenance: POMP-Pred: x12m; VCR x12m; MTX: x24m; 6-MPx24m.

ELIGIBILITY:
Inclusion Criteria:

* 14-55 years old;
* Ph-like ALL newly diagnosed;
* signed written informed consent

Exclusion Criteria:

* Pregnant women;
* History of pancreatitis;
* History of diabetes;
* History of active peptic ulcer disease in the past 6 months;
* History of arteriovenous thrombosis in the past 6 months;
* Severe active infection;
* Allergic to any drugs in PDT-Ph-like-ALL.

Ages: 14 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-02-14 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Event free survival | 3 years
  EFS of Ph-like ALL group

SECONDARY OUTCOMES:
Minimum residual disease after induction | 3 months
  MRD after 1 course
CR after Induction Therapy | 3 months
  CR rate of Ph-like group
Death in induction | 3 months
Adverse events | 3 years
  AE during PDT-Ph-like
Relapse | 3 years
  Relapse of Ph-like ALL
Relapse free survival | 3 years
  RFS
Overall survival | 3 years
  OS

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hematology, Nanfang Hospital, Guangzhou, Guangdong, China